CLINICAL TRIAL: NCT03519425
Title: A Pragmatic Randomised Study to Optimise Screening, Prevention and Care for Tuberculosis in Malawi
Acronym: PROSPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); London School of Hygiene and Tropical Medicine (Other); University of Liverpool (Other); McGill University (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 17-050
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Tuberculosis; Hiv; Tuberculosis, Pulmonary
Keywords: Tuberculosis; HIV; Randomised controlled trial; Africa; Public Health; Screening
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: A pragmatic open, three-arm individually-randomised controlled trial and economic evaluation
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Standard of care) (No Intervention): Participants will be directed to the clinic waiting area to be seen by facility health workers who will direct all further care without any further input from the study team. Available to facility health workers will be:
  * Routine HIV testing and counselling, provided by Facility HIV Testers using a rapid fingerprick kit-based algorithm.
  * Routine TB screening, with both sputum smear microscopy and Xpert MTB/Rif testing available onsite.
  * Routine linkage to the onsite HIV clinic, where patients are registered and assessed for initiation onto antiretroviral therapy by facility HIV Care Clinic health workers. Malawi guidelines recommend universal treatment for HIV. HIV Care Clinic health workers will additionally have access to TB screening tests as described above.
  * Routine linkage to the onsite TB clinic, where patients are registered and initiated onto anti-TB treatment. Malawi guidelines recommend universal HIV testing for all patients with confirmed TB.
- Group 2 (Optimised HIV screening and linkage to care) (Active Comparator): Participants will be directed to the study room located in a separate building. After identity validation participants will be offered a supervised HIV self-testing intervention. Participants will be given brief pre-test instructions and will be asked to self-test in a private area using the OraQuick 1/2 (OraSure Technologies) oral fluid HIV kit. Participants will be supported to read their HIV test result by study Research Assistants, and provided with confirmatory HIV testing by the trained Research Assistants.
  * HIV-positive participants will be supported by Research Assistants to register at the onsite HIV care clinic, and all further care (including TB screening) will be directed by facility health workers without any further study input.
  * HIV-negative participants will be referred to the clinic waiting area (with a copy of their HIV test results) to be seen by the facility health workers who will direct all further investigations without further study input.
  Interventions: Other: Optimised HIV screening and linkage to care
- Group 3 (Optimised HIV and TB screening and linkage to care) (Active Comparator): Participants will be directed to the Study Room. After identity validation, they will be offered the HIV self-testing and linkage intervention as described above for Group 2. Additionally, they will be offered a TB screening intervention comprising of:
  * A digital chest x-ray using the study MinXray unit.
  * Chest x-rays will be immediately classified by the CAD4TB software running on the MinXray unit laptop as either "high probability of TB", or "low probability of TB".
  * Participants whose chest x-rays have a low probability of TB will be referred to facility health workers (at either the onsite HIV care clinic if HIV-positive, or the clinic waiting area), with copies of their results for further routine care, and without further study input.
  * Participants whose chest x-ray x-ray show a high probability of TB will submit a single spot sputum sample for Xpert testing (done in the clinic). Those with confirmed TB will be linked to register at the onsite TB clinic.
  Interventions: Other: Optimised HIV screening and linkage to care; Other: Optimised tuberculosis screening and linkage to care

INTERVENTIONS:
Other: Optimised HIV screening and linkage to care — As described in group descriptions
  Arms: Group 2 (Optimised HIV screening and linkage to care); Group 3 (Optimised HIV and TB screening and linkage to care)
Other: Optimised tuberculosis screening and linkage to care — As described in group descriptions
  Arms: Group 3 (Optimised HIV and TB screening and linkage to care)

SUMMARY:
A pragmatic open, three-arm individually-randomised controlled trial and economic evaluation will be conducted in one primary health care centre in Blantyre, Malawi, where HIV and TB are major contributors to early mortality.

Participants will be adults with symptoms of tuberculosis (cough of any duration) attending the primary clinic with an acute care episode. We will exclude adults who have taken treatment for TB within the previous 6-months, who are taking isoniazid preventive therapy, who are not resident of Blantyre, or who plan to move out of Blantyre in the following 6-months.

Participants will be randomly allocated into one of three groups:

Group 1: Standard of care: Participants will be seen by facility health workers and receive clinician-directed screening for HIV and TB according to Malawi national guidelines.

Group 2: Optimised HIV testing and treatment linkage: Participants will be offered testing for HIV using rapid oral fluid kits by research assistants. Those with confirmed HIV infection will be linked to the HIV care clinic where facility healthworkers will screen for TB using standard sputum-based diagnostics.

Group 3: Optimised TB diagnosis, HIV screening and treatment linkage: Participants will receive a high-throughput and high-sensitivity TB screening intervention, in addition to the HIV testing intervention. This will comprise of an initial digital chest x-ray classified by the CAD4TB image-recognition software as either "high probability of TB", or "low probability of TB". Participants whose x-rays are suggestive of TB will receive confirmatory sputum testing with Xpert MTB/Rif Ultra cartridges, whilst participants whose x-rays have a low probability of TB will be referred to facility healthworkers for routine care.

All participants will be seen at the health facility at day 56, where they will be tested for HIV (if not on ART) and screened for TB.

The Primary Trial Outcome will compare between groups the time to tuberculosis treatment initiation by day 56. The trial is sufficiently powered to permit 3 pairwise comparisons between groups (i.e. Group 1 vs. 2; Group 2 vs. 3; and Group 1 vs. 3).

This three-arm pragmatic trial design allows us to efficiently answer two separate, important public health questions: firstly, by comparing Group 2 to Group 1, we should be able to determine whether HIV care should be prioritised for adults with TB symptoms. Additionally, by comparing Group 3 to Group 2, we will provide strong evidence for the effectiveness of an optimised and integrated HIV and TB diagnostic and treatment linkage approach.

DETAILED DESCRIPTION:
Ambitious global targets have been set to eliminate tuberculosis as a public health problem by 2035. However, in Africa, where HIV has driven extremely high incidence rates, progress in reducing new infections and TB deaths remains too slow.

We have previously demonstrated that adults seeking diagnosis and treatment for TB and HIV face considerable barriers, and have long delays in starting treatment with high pre-treatment mortality.

Efforts to reduce TB mortality have been hampered by limitations in TB diagnostics, with considerable uncertainty about how available and new tests can be best implemented.

The aim of the PROSPECT Study is therefore to investigate the effectiveness and cost-effectiveness of optimised TB/HIV diagnosis and treatment linkage interventions on TB and HIV case detection, treatment initiation and mortality.

Study design A pragmatic open, three-arm individually-randomised controlled trial and economic evaluation will be conducted in one primary health care centre in Blantyre, Malawi.

Study site and participants The study will be conducted at one primary health clinic in Blantyre Malawi, where we have established HIV and TB research facilities and previously demonstrated high need for improved TB and HIV diagnosis. Sputum-based TB diagnostics (smear microscopy, and Xpert MTB/Rif) and treatment, and comprehensive HIV care (including provider-initiated HIV testing and antiretroviral therapy) are available free-to-cost to patients through the Malawi national TB and HIV programmes.

Participants will be adults with symptoms of pulmonary tuberculosis (cough of any duration) attending the primary clinic with an acute care episode. We will exclude adults who have taken treatment for TB within the previous 6-months, or who are taking isoniazid preventive therapy, or who do not live in Blantyre, or plan to move out of Blantyre.

Interventions

Participants will be randomly allocated into one of three groups:

Group 1 - Standard of care: Participants will be seen by facility health workers and receive clinician-directed screening for HIV and TB according to Malawi national guidelines without further study input.

Group 2 - Optimised HIV testing and treatment linkage: Participants will be offered testing for HIV using rapid oral fluid kits by research assistants. Those with confirmed HIV infection will be linked to the HIV care clinic where facility healthworkers will screen for TB using standard sputum-based diagnostics without further study input.

Group 3 - Optimised TB diagnosis, HIV screening and treatment linkage: Participants will receive a high-throughput and high-sensitivity TB screening intervention, in addition to the HIV testing intervention. This will comprise of an initial digital chest x-ray classified by the CAD4TB image-recognition software as either "high probability of TB", or "low probability of TB". Participants whose x-rays are classified as having high probability of TB will receive confirmatory sputum testing with Xpert MTB/Rif cartridges, whilst participants whose x-rays have a low probability of TB will be referred to facility healthworkers for routine care.

All participants will be seen at the health facility at day 56, where they will be assessed to determine whether they are taking treatment for tuberculosis by inspection of medication, inspection of treatment cards, and inspection of facility TB registers. They will also be offered testing for HIV (if not on ART) and screened for TB, including by sputum culture, Xpert and smear microscopy.

Outcomes The primary trial outcome will be time in days - from Day 0 up to but not including Day 56 - to tuberculosis treatment initiation, evaluated at Day 56 following randomization. The trial is sufficiently powered to permit 3 pairwise comparisons between groups (i.e. Group 1 vs. 2; Group 2 vs. 3; and Group 1 vs. 3).

This three-arm pragmatic trial design allows us to efficiently answer two separate, important public health questions: firstly, by comparing Group 2 to Group 1, we should be able to determine whether HIV care should be prioritised for adults with TB symptoms. Additionally, by comparing Group 3 to Group 2, we will provide strong evidence for the effectiveness of an optimised and integrated HIV and TB diagnostic and treatment linkage approach.

Statistical considerations Assuming 17% of participants in Group 1 initiate TB treatment by 8-weeks, and 5% loss to-follow-up, a sample size of n=1455 participants randomised in a 1:1:1 ratio across the three groups provides at least 80% power to detect a hazard ratio of 1.5 comparing Group 2 to Group 1, and a hazard ratio of 1.41 comparing Group 3 to Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Attends Study Clinic with an acute care episode
* 18 years of age or older on the day of clinic attendance
* Has symptoms of tuberculosis (cough of any duration)
* Is resident within urban Blantyre
* Provides informed consent to participate

Exclusion Criteria:

* Taking treatment for tuberculosis on the day of clinic attendance
* Has taken any treatment for tuberculosis in the 6-months prior to clinic attendance
* Is taking isoniazid preventive therapy
* Plans to move out of Blantyre to live elsewhere in the following 6-months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1455 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Time to tuberculosis treatment initiation | Measured at 56 days after randomisation
  The primary trial outcome will be time in days - from Day 0 up to but not including Day 56 - to tuberculosis treatment initiation, evaluated at Day 56 following randomization.
  Analysis of the primary outcome will be done on an intention to treat basis, with all participants analysed according to the group to which they were randomised. Time to TB treatment outcome analysis will be right censored at Day 56 from randomisation if TB treatment is not initiated, or at day of loss to follow-up. We will make three pair-wise comparisons (Group 2 vs. Group 1; Group 3 vs. Group 2; and Group 3 vs. Group 1).

SECONDARY OUTCOMES:
Same day TB treatment initiation | Measured at 56 days after randomisation
  The proportion of randomised participants initiated onto tuberculosis treatment on the same day as randomisation, with the numerator being participants who were initiated on tuberculosis treatment on Day 0, and the denominator being all randomised participants.
Undiagnosed/untreated microbiologically-confirmed pulmonary tuberculosis | Measured at 56 days after randomisation
  The proportion of randomised participants with undiagnosed/untreated microbiologically-confirmed pulmonary TB at Day 56, with the numerator being participants with microbiologically-confirmed tuberculosis (either sputum culture, or sputum Xpert, or sputum smear microscopy positive on a sample taken on Day 56) and who are confirmed not to be taking tuberculosis treatment on Day 56 (including participants who have previously initiated tuberculosis treatment, but have defaulted or stopped treatment - regardless of reason - for at least one week). The denominator will be all randomised participants.
Undiagnosed/untreated HIV | Measured at 56 days after randomisation
  The proportion of randomised participants with undiagnosed/untreated HIV at Day 56, with the numerator being participants with positive confirmatory HIV test results at Day 56 and who are not taking antiretroviral therapy (regardless of previous HIV test results during or before the study period), and the denominator being all randomised participants.
Time to antiretroviral therapy initiation | Measured at 56 days after randomisation
  Time in days - from Day 0 up to but not including Day 56 - to initiation of antiretroviral therapy among participants with positive confirmatory HIV test results at Day 56 and who were not taking antiretroviral therapy at Day 0.
  Initiation of antiretroviral therapy will be defined by:
  A participant in whom there is documented evidence of commencement of combination antiretroviral therapy treatment, either by: inspection of the participant-carried national HIV programme treatment card; or inspection of the facility antiretroviral therapy treatment register; or inspection of antiretroviral therapy medication bottles or pill boxes.
Mortality | Measured at 56 days after randomisation
  The proportion of randomised participants reported to have died by Day 56, with the numerator being participants confirmed to have died through home tracing visits or TB treatment records, and the denominator being all randomised participants.
TB treatment outcome | Measured at 6-months after randomisation
  The proportion of TB cases with a successful TB treatment outcome. The numerator will be participants who were initiated onto tuberculosis treatment (either microbiologically-confirmed or clinically-diagnosed tuberculosis) up to, but not including Day 56, and who have a successful TB treatment outcome (either cured or completed treatment) at 6-months after starting treatment. The denominator will be all participants confirmed to have initiated tuberculosis treatment between Day 0 and up to, but not including Day 56.
Quality of life (EQ5D utility score) | Measured at 56 days after randomisation
  Mean difference in EuroQoL EQ5D utility score at Day 56, adjusting for participants' EQ5D utility score measured at Day 0.
Quality of life (EQ5D visual analogue scale) | Measured at 56 days after randomisation
  Mean difference in EuroQoL EQ5D visual analogue scale score, adjusting for participants' EQ5D visual analogue scale score measured at Day 0.
Cost-effectiveness | Measured at 56 days after randomisation
  Incremental cost-effectiveness per QALY gained

OTHER OUTCOMES:
Sex-and microbiological TB status-stratified analysis | Measured at 56 days after randomisation
  Although not statistically powered for comparison, in pre-specified exploratory sub-group analysis, we will stratify analysis of comparisons between pairs of groups for the primary outcome of time to tuberculosis treatment initiation (stratified by sex, and by microbiological TB status), and for the secondary outcomes of the proportion of participants with undiagnosed/untreated microbiologically-confirmed TB (stratified by sex), and undiagnosed/untreated HIV (stratified by sex).
  These pre-specified exploratory analyses will be done for hypothesis-generating purposes and to support the case for future research, as our previous studies have shown that men fare considerable worse than women throughout the TB and HIV diagnostic and care pathways.
Exploratory Bayesian analysis | Measured at 56 days after randomisation
  We will additionally undertake a Bayesian analysis of the primary trial outcome. Prior distributions for the proportion of participants initiating TB treatment will be elicited from key stakeholder groups, including community members, clinicians, researchers, TB experts, and policymakers.
  Key stakeholders will be invited to attend workshop meetings, where they will be introduced to the study design and interventions through presentations and group discussions. To elicit prior beliefs for effect of interventions, we will use a "bin-and-chip" method, implemented within an interactive web application.
  Using Bayes' theorem, we will combine elicited stakeholder group-specific log hazard ratio prior distributions with log-likelihood hazard ratio distributions from each pairwise comparison being made in the PROSPECT Study to construct posterior probability distributions.

CONTACTS AND LOCATIONS:
Locations (1):
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Chichiri, Malawi

IPD SHARING:
Plan to Share IPD: Yes
We are strongly committed to ensuring that the trial datasets are made openly available, and that all code used in the analysis are published to allow fully reproducible research. The data collected by this research will be of importance to other researchers and the public, and could for example be used by other researchers conducting meta-analysis, or by policymakers modelling the potential return on investment of implementing interventions within their settings.
  Therefore, we will establish a public online GitHub repository, where the final anonymised individual participant trial dataset and code to allow reproduction of all analysis will be published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within four months of trial completion
Access Criteria: Open access

REFERENCES:
- [Derived] MacPherson P, Webb EL, Kamchedzera W, Joekes E, Mjoli G, Lalloo DG, Divala TH, Choko AT, Burke RM, Maheswaran H, Pai M, Squire SB, Nliwasa M, Corbett EL. Computer-aided X-ray screening for tuberculosis and HIV testing among adults with cough in Malawi (the PROSPECT study): A randomised trial and cost-effectiveness analysis. PLoS Med. 2021 Sep 9;18(9):e1003752. doi: 10.1371/journal.pmed.1003752. eCollection 2021 Sep. PMID 34499665
- [Derived] MacPherson P, Webb EL, Lalloo DG, Nliwasa M, Maheswaran H, Joekes E, Phiri D, Squire B, Pai M, Corbett EL. Design and protocol for a pragmatic randomised study to optimise screening, prevention and care for tuberculosis and HIV in Malawi (PROSPECT Study). Wellcome Open Res. 2018 Nov 21;3:61. doi: 10.12688/wellcomeopenres.14598.3. eCollection 2018. PMID 30542662